CLINICAL TRIAL: NCT04399850
Title: Impact of Hypnosis During Invasive Procedure in Intensive Care Unit
Acronym: HYPNOICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: APHP191042
Record Dates: First submitted 2020-04-29; First posted 2020-05-22 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Pain
Keywords: invasive procedure; pain distress; hypnosis
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who receive hypnosis (Experimental): Patients who receive hypnosis during procedure by experiment physician
  Interventions: Other: Hypnosis group
- Control arm (No Intervention): Patient with conventional pain management

INTERVENTIONS:
Other: Hypnosis group — Patients who receive hypnosis
  Arms: Patients who receive hypnosis

SUMMARY:
Pain during ICU stay remains one of the major complaints for patients. Beside pain intensity, well described by patients' self reports, pain distress, which is an emotional experience, cannot be treated with usual analgesia. The aim of the study is to analyze the impact of hypnosis on pain intensity and distress on short and long term outcomes in non-sedated ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years and older
* ICU hospitalisation
* Non-sedated patients who need an invasive procedure (Invasive procedures are defined as chest tube (insert or remove), fibroscopy, catheter insert, lumbar punction and bone marrow aspiration)
* Physician experienced in hypnosis available
* written informed consent
* health insurance

Exclusion Criteria:

* sedation and intubation, delirium, end-of-life decision,
* deaf patient,
* patient who does not understand French language,
* pregnancy
* patient under guardianship or curatorship
* lack of health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Pain distress | within the before and the first hour after the procedure
  Pain distress change in the hypnosis group measured before and within the first hour after the procedure.
  Pain distress will be assessed using Numeric rating scale, which goes from 0 (no pain stress) to 10 (maximum pain stress).

SECONDARY OUTCOMES:
Pain intensity | within first hour and first 24 hours after procedure
  Pain intensity will be assessed using Numeric rating scale, which goes from 0 (no pain) to 10 (maximum pain imaginable).
Number of adverse events | during procedure
Length of each painful procedure | up to 3 months
Analgesia dose | within first and 24 hours after procedure
  The dose of each analgesia treatment received by the patient will be collected.
Type of analgesia | within first and 24 hours after procedure
  The type of each analgesia treatment received by the patient will be collected.
Anxiety | within first and 24 hours after procedure
  Anxiety within first and 24 hours after procedure will be assessed using Numeric rating scale, which goes from 0 (no anxiety) to 10 (maximum anxiety imaginable).
Hospital Anxiety and Depression (HAD) scale | at 3 months
  The HAD scale is a self-assessment scale for detecting states of depression and anxiety in the setting of an hospital medical outpatient clinic.
  HAD scale is a self-administered scale of 14 items which assessed levels of depression and anxiety, divided into 2 subscales of 7 items (Anxiety or HADS-A, Depression or HADS-D). Each item is scored on a scale of 0 to 3. A score is generated for each of the two sub-scales (sum of the 7 items, ranging from 0 to 21). A higher score indicates worse outcome.
Post traumatic stress disorder assessed using Impact of Event Scale Revisited (IES R) | at 3 months
  The IES-R is a 22-item self-report measure (for DSM-IV) that assesses subjective distress caused by traumatic events. Items are rated on a 5-point scale ranging from 0 to 4 . The IES-R yields a total score (ranging from 0 to 88)
Proportion of patients who had hypnosis transe | during procedure
Description of the experience of hypnosis | at 3 months
  Qualitative analysis of the experience of hypnosis will be performed using the semi-structured interview

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint-Louis, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided